CLINICAL TRIAL: NCT01072968
Title: Efficacy and Safety of BF2.649 in Treatment of Excessive Daytime Sleepiness in Patients With Obstructive Sleep Apnea (OSA) Refusing the Nasal Continuous Positive Airway Pressure (nCPAP) Therapy
Brief Title: BF2.649 in Patients With OSA, Still Complaining of EDS and Refusing to be Treated by CPAP.
Acronym: HAROSA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P09-09 / BF2.649
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Obstructive Sleep Apnea; Excessive Daytime Sleepiness
Keywords: Multicenter; Randomized; Double-blind; Efficacy and safety study; BF2.649 versus placebo; Patients suffering from Obstructive Sleep Apnea; Complaining from Excessive Daytime Sleepiness; Refusing nasal Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BF2.649 (Experimental): BF2.649 capsules dosed at 5 mg, 10 mg, 20 mg
  Interventions: Drug: BF2.649
- Placebo (Placebo Comparator): Capsules of placebo containing lactose with low, medium and high dosage
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BF2.649 — 1 capsule per day in the morning before the breakfast
  Other Names: Pitolisant
  Arms: BF2.649
Drug: Placebo — 1 capsule per day in the morning before the breakfast
  Arms: Placebo

SUMMARY:
Multicenter randomized double blind study versus placebo during 12 weeks with at first, an escalating dose period followed by stable dose period at the selected dose.

This double-blind period can be followed by a 9 months open-label period if the patient wishes to continue with the study product.

DETAILED DESCRIPTION:
The first period (12 weeks double blind period) will aim at demonstrating the efficacy and safety of BF2.649 by verifying whether the results of BF2.649 are superior to those of placebo.

The aim of the second period (open label extension phase) will be to assess the long-term tolerance, as well as the maintenance of the BF2.649 efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OSA still complaining EDS,refusing nCPAP
* ESS score ≥ 12

Exclusion Criteria:

* Patients suffering from insomnia without OSA
* Co-existing narcolepsy
* Patient with sleep debt not due to OSA
* Acute or chronic severe disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
ESS (Epworth Sleepiness Scale) change from baseline | From baseline to week 12 and week 51

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne De Paillette, MD, Study Director — Bioprojet
Locations (1):
- Centre Hospitalier Universitaire de Grenoble, Grenoble, Grenoble, France

REFERENCES:
- [Derived] Pepin JL, Attali V, Causse C, Verbraecken J, Hedner J, Lecomte I, Tamisier R, Levy P, Lehert P, Dauvilliers Y. Long-Term Efficacy and Safety of Pitolisant for Residual Sleepiness Due to OSA. Chest. 2024 Mar;165(3):692-703. doi: 10.1016/j.chest.2023.11.017. Epub 2023 Nov 17. PMID 37979718
- [Derived] Dauvilliers Y, Verbraecken J, Partinen M, Hedner J, Saaresranta T, Georgiev O, Tiholov R, Lecomte I, Tamisier R, Levy P, Scart-Gres C, Lecomte JM, Schwartz JC, Pepin JL; HAROSA II Study Group collaborators. Pitolisant for Daytime Sleepiness in Patients with Obstructive Sleep Apnea Who Refuse Continuous Positive Airway Pressure Treatment. A Randomized Trial. Am J Respir Crit Care Med. 2020 May 1;201(9):1135-1145. doi: 10.1164/rccm.201907-1284OC. PMID 31917607